CLINICAL TRIAL: NCT02838940
Title: Preventive Antibiotic Serum Levels During Caesarean Section
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0147-16-TLV
Record Dates: First submitted 2016-05-29; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Blood Antibiotic Levels
MeSH Terms: interventions — Blood Specimen Collection; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cesarean in different indications (Experimental): Women that are about to undergo an elective cesarean in different indications.
  Interventions: Procedure: Blood samples.; Drug: Cefazolin

INTERVENTIONS:
Procedure: Blood samples. — At the beginning of the first incision in the skin, first blood sample will be taken for levels of antibiotics in serum test.
  Second blood sample for drug levels in serum test, will be taken while closing the surgical incision in the skin at the end of the operation.
Drug: Cefazolin — According to the ward protocol prior to the anesthesia by an anesthesiologist, the women will receive one dose of 1 g Cefazolin the usual loading dose. Women with a BMI over 30 will receive Cefazolin of about 2 grams.

SUMMARY:
Background

Preventive antibiotic treatment before performing invasive procedures is a basic element in preventing infections. The essence of preventive antibiotic treatment is strengthening the defense mechanisms of the immune system by preserving a certain drug levels in the blood. The timing of giving the antibiotics is very important. Several research groups have tried to check the levels of Cefazolin (the most common antibiotics in the field of obstetrics) in serum and adipose tissue in women during cesarean. These groups presented conflicting research results.

OBJECTIVE

This study will discuss the preventive antibiotic treatment levels accepted prior cesareans, to determine:

1. What are the factors affecting the level of drug in the blood?
2. Is there a fixed time which beyond it, blood drug levels are below the MIC(Minimal Inhibitory Concentration)?
3. Is the provision of usual preventive care also addresses the situations of metabolic disorder?

DETAILED DESCRIPTION:
Background

Preventive antibiotic treatment before performing invasive procedures is a basic element in preventing infections. The essence of preventive antibiotic treatment is strengthening the defense mechanisms of the immune system by preserving a certain drug levels in the blood. The timing of giving the antibiotics is very important. Several research groups have tried to check the levels of Cefazolin (the most common antibiotics in the field of obstetrics) in serum and adipose tissue in women during cesarean. These groups presented conflicting research results.

OBJECTIVE

This study will discuss the preventive antibiotic treatment levels accepted prior cesareans, to determine:

1. What are the factors affecting the level of drug in the blood?
2. Is there a fixed time which beyond it, blood drug levels are below the MIC(Minimal Inhibitory Concentration)?
3. Is the provision of usual preventive care also addresses the situations of metabolic disorder?

PATIENTS & METHODS

Women that meet the inclusion criteria and are about to undergo cesarean in different indications, in elective and urgent way.

1. Before performing TIMEOUT outside the surgery room, The investigators will explanation about the process and purpose of the study, and informed consent will be obtained.
2. Prior to the anesthesia by an anesthesiologist, the women will receive one dose of 1 g Cefazolin the usual loading dose. Women with a BMI over 30 will receive Cefazolin of about 2 grams.
3. With the beginning of the first incision in the skin, first blood sample will be taken to test levels of antibiotics in serum.
4. Second blood sample to test drug levels in serum will be taken while closing the surgical incision in the skin at the end of the operation.
5. The continuation of post surgery recovery process will be as usual, in accordance with departmental protocols.

With the results of tissue and serum samples, segmentation which compares the drug levels in the different tissues will be performed.Also, the correlation between drug levels in women with different BMI and morbidities that may cause measurable or not pharmacokinetic changes will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of 37 weeks and above.
2. Women who arrive to elective cesareans.
3. Age of women: 18-50 years old.

Exclusion Criteria:

1. Suspected clinical / laboratory active infection
2. urgent surgery
3. Sensitivity to penicillin or cephalosporins antibiotics that requires antibiotics change.
4. Women who received the week before surgery antibiotic treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Blood antibiotic levels | 30 min- 2 hours.
  Blood MIC(Minimal Inhibitory Concentration) levels of antibiotic will be checked at first incision and at the time of closing surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No